CLINICAL TRIAL: NCT01550055
Title: CMAB009 Plus Irinotecan Versus Irinotecan-only as Second-line Treatment After Fluoropyrimidine and Oxaliplatin Failure in KRAS Wild-type Metastatic Colorectal Cancer Patients: Prospective, Open-label, Randomized, Phase II/III Trial
Brief Title: Study of CMAB009 to Treat KRAS Wild Type Metastatic Colorectal Cancer
Acronym: CRC009
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shanghai Zhangjiang Biotechnology Limited Company (Industry)
Collaborators: Shanghai Biomabs Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMAB009mCRCⅡ/Ⅲ; CMAB009 (Registry Identifier: 2007L02499)
Record Dates: First submitted 2012-03-07; First posted 2012-03-09 (Estimated); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Metastatic Colorectal Cancer
Keywords: KRAS wild-type; Metastatic Colorectal Cancer; CMAB009 Plus Irinotecan; Phase II/III
MeSH Terms: conditions — Colorectal Neoplasms | interventions — CMAB009; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CMAB009 plus Irinotecan (Experimental)
  Interventions: Drug: CMAB009 plus Irinotecan
- Irinotecan-only and sequential-CMAB009 (Active Comparator)
  Interventions: Drug: Irinotecan-only and sequential-CMAB009

INTERVENTIONS:
Drug: CMAB009 plus Irinotecan — Combined with irinotecan 180 mg/m2 every 2 weeks, CMAB009 400 mg/m2 day 1 followed by 250 mg/m2 weekly till disease progression
  Other Names: YiMaiLin for irinotecan
  Arms: CMAB009 plus Irinotecan
Drug: Irinotecan-only and sequential-CMAB009 — First, irinotecan 180 mg/m2 every 2 weeks till PD occured, discontinue it; then, CMAB009 400 mg/m2 day 1 followed by 250 mg/m2 weekly till disease progression.
  Other Names: YiMaiLin for irinotecan
  Arms: Irinotecan-only and sequential-CMAB009

SUMMARY:
The primary purpose of this study is to evaluate the clinical response and safety of CMAB009 plus irinotecan versus irinotecan-only as second-line treatment after fluoropyrimidine and oxaliplatin failure in KRAS wild-type metastatic colorectal cancer patients

DETAILED DESCRIPTION:
CMAB009 is a recombinant, human/mouse chimeric monoclonal antibody (mAb) that binds specifically to the extracellular domain of EGFR. It is composed of the Fv regions of a murine anti-EGFR antibody with human IgG1 heavy and k light chain constant regions and it is expressed by Chinese hamster ovary cells. It has the same amino acid sequence as cetuximab (C225, Erbitux®) , but it has slightly different abilities for glycosylation and other post-translational modifications, and it is developed by Shanghai Zhangjiang Biotechnology Limited Company and produced by Biomabs. Phase I study results suggest that CMAB009 showed well-tolerated safety profile and primary efficacy. This multicenter, open-label study was to determine whether adding CMAB009 to irinotecan increased the response rate and prolongs survival in patients with KRAS wild-type metastatic colorectal cancer (mCRC) previously treated with fluoropyrimidine and oxaliplatin.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed metastatic colorectal adenocarcinoma
* KRAS wild-type tumors, EGFR-expressing or EGFR-nonexpressing by immunohistochemistry;
* has measurable lesion, at least 1cm in diametre by CT or MRI, at least 2cm diametre by physical examination or other iconography
* ECOG performance status 0 to 1
* Failure (disease progression/discontinuation due to toxicity) of fluoropyrimidine and oxaliplatin treatment,stop at least one month thereafter, irinotecan-naïve

Exclusion Criteria:

* Previous irinotecan or anti-EGFR therapies
* hematologic function: hemoglobin, less than 90g per liter; neutrophil count, less than 1500 per cubic millimeter; and platelet count, less than 100,000 per cubic millimeter
* liver function: bilirubin, more than 1.0 times the upper limit of normal; aspartate aminotransferase and alanine aminotransferase, more than 5.0 times and 2.5 times the upper limit of normal with hepatic metastasis or not
* Renal function: serum creatinine, more than 1.5 times the upper limit of normal
* Patients with symptomatic central nervous system metastases

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 512 (Actual)
Dates: Start 2009-05-31 (Actual); Primary Completion 2012-12-23 (Actual); Study Completion 2015-07-23 (Actual)

PRIMARY OUTCOMES:
Overall response rate | Time to progression, assessed up to two years
  Tumor response was evaluated every 6 weeks and confirmed at least 4 weeks later

SECONDARY OUTCOMES:
Progression-free Survival | Time to progression, assessed up to two years
  The study was designed to evaluate the PFS as second end point, progression-free survival is defined as the period from date of randomization to date of disease progression

CONTACTS AND LOCATIONS:
Overall Officials: Yuankai Shi, M.D., Study Chair — Cancer Institute and Hospital, Chinese Academy of Medical Sciences; B C Mei, Principal Investigator — Peking Union Medical College Hospital; B Li, Principal Investigator — Chinese PLA Affiliated Central Hospital; X J Ming, Principal Investigator — Affiliated Hospital of Chinese PLA Military Academy of Medical Science; B Yi, Principal Investigator — TianJin Medical University Affiliated Cancer Hospital; Y Qiang, Principal Investigator — NanKai University Affiliated Hospital; L Wei, Principal Investigator — HeBei Medical University Fouth Hospital; L Y Peng, Principal Investigator — Chinese Medical University First Affiliated Hospital; W B Cheng, Principal Investigator — Jinan Military Central Hospital; W Z Hai, Principal Investigator — Shandong Provincal Cancer Hospital; Y S Ying, Principal Investigator — Tongji Medical College of Huazhong University of Science and Technology; L Yi, Principal Investigator — Hunan Provincal Cancer Hospital; C Y Gui, Principal Investigator — Fujian Provincal Cancer Hospital; W L Wei, Principal Investigator — Shanghai Jiaotong University Affiliated First People's Hospital; Z Jun, Principal Investigator — Shanghai Jiaotong University Affiliated Ruijin Hospital; H C Hong, Principal Investigator — Central South University; OY Xuenong, Principal Investigator — Fuzhou Central Hospital of Nanjing Military Command; L Jin, Principal Investigator — Fudan University Affiliated Cancer Hospital; Z Y Ping, Principal Investigator — Zhejiang Provincal Cancer Hospital; H X Hua, Principal Investigator — Guangxi Medical University Affiliated Cancer Hospital; L R Cheng, Principal Investigator — Nanfang Medical University Affiliated Nanfang Hospital; L Y Hong, Principal Investigator — Zhongshan University Affliated Cancer Hospital; T Min, Principal Investigator — Suzhou University Affiliated First Hospital; Z Z Xiang, Principal Investigator — Suzhou University Affiliated Second Hospital; C Ying, Principal Investigator — Jilin Provincal Cancer Hospital; F J Feng, Principal Investigator — Jiangsu Provincal Cancer Hospital; Q S Qui, Principal Investigator — Chinese PLA Affiliated 81 Hospital; J Bin, Principal Investigator — Shanghai Jiaotong University Affiliated Third People's Hospital; Z R Sheng, Principal Investigator — The First Affiliated Hospital of Bengbu Medical University; M G Xin, Principal Investigator — Nantong Medical College Affiliated Hospital; S G Ping, Principal Investigator — Anhui Medical University Affiliated First Hospital; D W Chao, Principal Investigator — The Fourth Military University Affiliated First Hospital; L H Jie, Principal Investigator — The Third Military University Affiliated First Hospital; X Ying, Principal Investigator — Chongqing University Cancer Hospital; F Min, Principal Investigator — Chongqing First People's Hospital; B Feng, Principal Investigator — Sichuan University Huaxi Hospital; W D Lin, Principal Investigator — Sichuan Provincal People's Hospital; Z W Hua, Principal Investigator — Gansu Provincal Cancer Hospital; C Hong, Principal Investigator — Kunming Central Hospital of Chengdu Military Command

REFERENCES:
- [Derived] Shi Y, Li J, Xu J, Sun Y, Wang L, Cheng Y, Liu W, Sun G, Chen Y, Bai L, Zhang Y, He X, Luo Y, Wang Z, Liu Y, Yao Q, Li Y, Qin S, Hu X, Bi F, Zheng R, Ouyang X. CMAB009 plus irinotecan versus irinotecan-only as second-line treatment after fluoropyrimidine and oxaliplatin failure in KRAS wild-type metastatic colorectal cancer patients: promising findings from a prospective, open-label, randomized, phase III trial. Cancer Commun (Lond). 2019 May 24;39(1):28. doi: 10.1186/s40880-019-0374-8. PMID 31126331